CLINICAL TRIAL: NCT04475666
Title: Replacing Protein Via Enteral Nutrition in a Stepwise Approach in Critically Ill Patients: An International, Multicenter Randomized Controlled Trial
Brief Title: Replacing Protein Via Enteral Nutrition in Critically Ill Patients
Acronym: REPLENISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC19/414/R
Record Dates: First submitted 2020-06-07; First posted 2020-07-17 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness; Nutrition Disorders
MeSH Terms: conditions — Critical Illness; Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Replenish protein group (Active Comparator): The subjects randomized to this group will receive the standard amount of proteins (maximum 1.2 g/kg/day) from the primary polymeric formula AND supplemental protein at 1.2 g/kg/day
  Interventions: Other: Replenish protein group
- Standard protein group (Active Comparator): The subjects randomized to this group will receive standard prescription without supplemental proteins (maximum1.2 g/kg/day) from the primary polymeric formula. No supplemental protein will be allowed
  Interventions: Other: Standard protein group

INTERVENTIONS:
Other: Replenish protein group — For patients with Body mass index(BMI) <30, use pre-ICU actual body weight(BW) for the calculation; if unavailable, use weight on ICU admission. For patients with BMI >=30, use adjusted body weight
  Arms: Replenish protein group
Other: Standard protein group — For patients with BMI <30, use pre-ICU actual BW for the calculation; if unavailable, use weight on ICU admission. For patients with BMI >=30, use adjusted body weight
  Arms: Standard protein group

SUMMARY:
The investigator will investigate the effect of supplemental enteral protein (1.2 g/kg/day) added to standard formula to achieve high amount of enteral protein (range 2-2.4 g/kg/day) given from ICU day 5 until ICU discharge up to ICU day 90 as compared to no supplemental enteral protein to achieve moderate amount enteral protein (0.8-1.2 g/kg/day), given in conjunction with similar amounts of stepwise caloric administration in the two groups on all-cause 90-day mortality.

DETAILED DESCRIPTION:
The REPLENISH is a multicentric, international, open label, randomized controlled trial which will enroll subjects in intensive care unit. Patients will be randomized on day 4 of ICU admission. Until ICU day 4, protein requirement will be provided according to the local practice as long as no intravenous amino acids are given and the average protein intake in the first 4 days does not exceed 0.8 g/kg/day. On ICU day 4, patients will be randomized to one of the two treatment groups: one with standard prescription without supplemental proteins (maximum1.2 g/kg/day) from the primary polymeric formula and another group will receive the standard amount of proteins (maximum 1.2 g/kg/day) from the primary polymeric formula AND supplemental protein at 1.2 g/kg/day.

Randomization will be stratified by suspected COVID-19 and then by site and the use of renal replacement therapy at the time of randomization (intermittent hemodialysis or continuous renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria(on ICU calendar day 4 or the morning of day 5)

1. Age ≥18-years old
2. Patient started on enteral nutrition (EN) via nasogastric/orogastric or duodenal or percutaneous endoscopic gastrostomy (PEG) or jejunostomy tubes.
3. The patient is on invasive mechanical ventilation and unlikely to be discharged from ICU next day.

Exclusion Criteria:

1. Lack of commitment to full life support or brain death. Patients with "Do Not Resuscitate" order but with commitment to ongoing life support can be enrolled.
2. Patients on any amount of parenteral nutrition (PN) in ICU at the time of screening, whether PN is used alone or in combination with enteral nutrition. Non-nutritional calories (dextrose, propofol, citrate) not considered as PN.
3. Patients who received an average protein of more than 0.8g/kg/day in the first 4 ICU days.
4. Patients being fed entirely through oral route - i.e. those who are eating.
5. Pregnancy.
6. Burn patients.
7. Prisoners or those undergoing forced treatment.
8. Patients with hepatic encephalopathy or Child C liver cirrhosis
9. Inherited defect of amino acid metabolism.
10. Allergies to protein supplement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2502 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
90 day-all cause mortality | 90 days
  Mortality 90 days post randomization

SECONDARY OUTCOMES:
Days alive at day 90 without life support | 90 days
  use of vasopressor/inotropic support, invasive mechanical ventilation and/or renal replacement therapy
Days alive and out of hospital at day 90 | 90 days
  90 day survival after randomization
Bacteremia until 2 days of ICU stay | until 2 days post ICU.
  Any symptoms of bacteremia
New or progression of Skin Pressure Ulcers | ICU stay
  anytime during ICU stay
Functional assessment at day 90 | Day 90
  SARC-F screen for sarcopenia and EuroQoL

OTHER OUTCOMES:
Safety outcomes during ICU stay | ICU stay
  New episode of stage 2 or higher AKI by KDIGO criteria; 2. Pneumonia defined as episodes of newly confirmed pneumonia according to the modified CDC criteria; 3. Grade IV Acute Gastrointestinal injury (AGI)
Minor safety outcomes during ICU stay | ICU stay
  Feeding tolerance; Diarrhoea; Refeeding syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Yaseen M Arabi, MD, Principal Investigator — King Saud Bin Abdulaziz University for Health Sciences
Locations (2):
- Saudi Arabia (2):
  - King Abdulaziz Medical city, Jeddah, Jeddah
  - Intensive Care Unit, King Abdulaziz Medical City, Riyadh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arabi YM, Casaer MP, Chapman M, Heyland DK, Ichai C, Marik PE, Martindale RG, McClave SA, Preiser JC, Reignier J, Rice TW, Van den Berghe G, van Zanten ARH, Weijs PJM. The intensive care medicine research agenda in nutrition and metabolism. Intensive Care Med. 2017 Sep;43(9):1239-1256. doi: 10.1007/s00134-017-4711-6. Epub 2017 Apr 3. PMID 28374096
- [Background] Liebau F, Wernerman J, van Loon LJ, Rooyackers O. Effect of initiating enteral protein feeding on whole-body protein turnover in critically ill patients. Am J Clin Nutr. 2015 Mar;101(3):549-57. doi: 10.3945/ajcn.114.091934. Epub 2015 Feb 4. PMID 25733640
- [Background] McClave SA, Taylor BE, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society for Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):159-211. doi: 10.1177/0148607115621863. No abstract available. PMID 26773077
- [Background] Compher C, Chittams J, Sammarco T, Nicolo M, Heyland DK. Greater Protein and Energy Intake May Be Associated With Improved Mortality in Higher Risk Critically Ill Patients: A Multicenter, Multinational Observational Study. Crit Care Med. 2017 Feb;45(2):156-163. doi: 10.1097/CCM.0000000000002083. PMID 28098623
- [Background] Weijs PJ, Looijaard WG, Beishuizen A, Girbes AR, Oudemans-van Straaten HM. Early high protein intake is associated with low mortality and energy overfeeding with high mortality in non-septic mechanically ventilated critically ill patients. Crit Care. 2014 Dec 14;18(6):701. doi: 10.1186/s13054-014-0701-z. PMID 25499096
- [Background] Koekkoek WACK, van Setten CHC, Olthof LE, Kars JCNH, van Zanten ARH. Timing of PROTein INtake and clinical outcomes of adult critically ill patients on prolonged mechanical VENTilation: The PROTINVENT retrospective study. Clin Nutr. 2019 Apr;38(2):883-890. doi: 10.1016/j.clnu.2018.02.012. Epub 2018 Feb 17. PMID 29486907
- [Background] Arabi YM, Aldawood AS, Al-Dorzi HM, Tamim HM, Haddad SH, Jones G, McIntyre L, Solaiman O, Sakkijha MH, Sadat M, Mundekkadan S, Kumar A, Bagshaw SM, Mehta S; PermiT trial group. Permissive Underfeeding or Standard Enteral Feeding in High- and Low-Nutritional-Risk Critically Ill Adults. Post Hoc Analysis of the PermiT Trial. Am J Respir Crit Care Med. 2017 Mar 1;195(5):652-662. doi: 10.1164/rccm.201605-1012OC. PMID 27589411
- [Background] Heyland DK, Patel J, Bear D, Sacks G, Nixdorf H, Dolan J, Aloupis M, Licastro K, Jovanovic V, Rice TW, Compher C. The Effect of Higher Protein Dosing in Critically Ill Patients: A Multicenter Registry-Based Randomized Trial: The EFFORT Trial. JPEN J Parenter Enteral Nutr. 2019 Mar;43(3):326-334. doi: 10.1002/jpen.1449. Epub 2018 Sep 27. PMID 30260486
- [Derived] Arabi YM, Al-Dorzi HM, Aldibaasi O, Sadat M, Jose J, Muharib D, Algethamy H, Al-Fares AA, Al-Hameed F, Mady A, Kharaba A, Al Bshabshe A, Maghrabi K, AlGhamdi K, Rasool G, AlGhamdi A, Almekhlafi GA, Chalabi J, AlHumedi HI, Sakkijha MH, Alamrey NK, Alaskar AS, Alhutail RH, Sifaoui K, Alqahtani R, Qureshi AS, Hejazi MM, Arishi H, AlQahtani S, Ghazi AM, Baaziz ST, Azhar AO, Alabbas SF, AlAqeely M, AlOrabi O, Al-Mutawa A, AlOtaibi M, Elghannam MF, Almaani M, Buabbas SF, Alfilfil WAM, Alshahrani MS, Starkopf J, Preiser JC, Perner A, AlMubarak JH, Hazem WM, Albrahim T, Al-Dawood A; and the Saudi Critical Care Trials Group. Statistical analysis plan for the replacing protein via enteral nutrition in a stepwise approach in critically ill patients (REPLENISH) randomized clinical trial. Trials. 2024 May 2;25(1):296. doi: 10.1186/s13063-024-08105-w. PMID 38698442
- [Derived] Arabi YM, Al-Dorzi HM, Sadat M, Muharib D, Algethamy H, Al-Hameed F, Mady A, AlGhamdi A, Almekhlafi GA, Al-Fares AA, Kharaba A, Al Bshabshe A, Maghrabi K, Al Ghamdi K, Rasool G, Chalabi J, AlHumedi HI, Sakkijha MH, Alamrey NK, Alhutail RH, Sifaoui K, Almaani M, Alqahtani R, Qureshi AS, Hejazi MM, Arishi H, AlQahtani S, Ghazi AM, Baaziz ST, Azhar AO, Alabbas SF, AlAqeely M, AlOrabi O, Al-Mutawa A, AlOtaibi M, Aldibaasi O, Jose J, Starkopf J, Preiser JC, Perner A, Al-Dawood A; Saudi Critical Care Trials Group. Replacing protein via enteral nutrition in a stepwise approach in critically ill patients: the REPLENISH randomized clinical trial protocol. Trials. 2023 Jul 30;24(1):485. doi: 10.1186/s13063-023-07507-6. PMID 37518058
- [Derived] Al-Dorzi HM, Stapleton RD, Arabi YM. Nutrition priorities in obese critically ill patients. Curr Opin Clin Nutr Metab Care. 2022 Mar 1;25(2):99-109. doi: 10.1097/MCO.0000000000000803. PMID 34930871